CLINICAL TRIAL: NCT00568490
Title: Identification of Secreted Markers for Tumor Hypoxia in Patients With Head and Neck or Lung Cancers
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB-10564; 73995 (Other: Stanford University Alternate IRB Approval Number); SU-11052007-801 (Other: Stanford University); R01DE029672-01A1 (NIH); NCT00185822 (obsolete NCT alias)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Lung Cancer; Lip Cancer; Lip Neoplasms; Head and Neck Cancers
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Lip Neoplasms | interventions — Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, tumor tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tumor biopsy — For patients who undergo tumor biopsy or resection at Stanford, approximately 500 mg of the tumor will be removed from the resection specimen
Procedure: Phlebotomy — Blood draw (approximately 20 cc) prior to any anticancer therapy Weekly blood draw (approximately 20cc) only for patients who are undergoing radiation treatment at Stanford University
  Other Names: Blood draw

SUMMARY:
The purpose of this study is to identify and confirm new blood and tissue markers for prognosis and tumor hypoxia. Tumor hypoxia, or the condition of low oxygen in the tumor, has been shown to increase the risk of tumor spread and enhance tumor resistance to the standard treatment of radiation and chemotherapy in head and neck and lung cancers. We have recently identified several proteins or markers in the blood and in tumors (including osteopontin, lysyl oxidase, macrophage inhibiting factor and proteomic technology) in the laboratory that may be able to identify tumors with low oxygen levels or more aggressive behaving tumors.

DETAILED DESCRIPTION:
The endpoints of the study are

1. To validate the prognostic significance of OPN in H&N and lung cancer patients and to monitor its level during active therapy and follow up for cancer surveillance.
2. To identify a gene and protein signature for hypoxia in H&N and lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck sites or non-small cell lung cancer, or relatives of patients with histologically confirmed squamous cell carcinoma of the head and neck.
* Able to sign a Stanford IRB approved consent form

Exclusion criteria:

* Refuse or unable to sign an IRB approved consent form.
* Refuse to be contacted in the future for follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 1998-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Identification of Secreted Markers for Tumor Hypoxia through tissue collection | before therapy, weekly during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States